CLINICAL TRIAL: NCT07063433
Title: The Effect of Gluma and Bioactive Glass in Treatment of Dentin Hypersensitivity in Cervical Lesions (A Randomized Clinical Trial)
Brief Title: Effect of Gluma and Bioactive Glass Desensitizers in Treatment of Dentin Hypersensitivity in Cervical Non-Carious Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Sara Katarya, Principal Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-012
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Dentin Hypersensitivity
Keywords: dentin hypersensitivity; gluma; Bioactive glass; fluoride varnish; VAS; non carious lesions; cervical non carious lesions
MeSH Terms: conditions — Dentin Sensitivity | interventions — gluma desensitizer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Gluma Group (Active Comparator): Each sensitive tooth will be cleaned with a polishing paste, rinsed with water and air dried. Two coats of Gluma Desensitizer will be applied using a disposable brush applicator following the manufacturer's instructions and left untouched for 30-60 minutes.
  Interventions: Drug: Gluma Desensitizer
- Bioactive Glass Group (Active Comparator): To maintain a dry and clear field of vision, cheek retractors and high-volume suction will be employed during the procedure. High-volume suction, featuring a 45-degree beveled end, will be strategically positioned at the incisal or occlusal part of the teeth. This placement is designed to efficiently remove any particles, preventing the patient from swallowing them and minimizing the risk of minor injuries resulting from a forceful powder and water stream. The NSK Prophymate Neo will be utilized to dispense Sylc dry powder, which comprises calcium sodium phosphosilicate, onto the sensitive areas. The air stream will be carefully adjusted to 40-46 psi in accordance with the manufacturer's instructions. The handpiece will be maintained at a constant distance of 3-4 mm from the tooth surface, positioned at 60-80 degrees on the buccal surfaces. To prevent gingival injury, the tip of the handpiece will be directed incisally during application. The powder will be applied for 5-10 seconds pe
  Interventions: Drug: Bioactive glass
- Combination of Gluma and Bioactive glass (Active Comparator): A combination of both Gluma and bioactive glass powder will be applied to the assigned teeth.
  Interventions: Drug: Gluma Desensitizer; Drug: Bioactive glass
- Fluoride Varnish (Active Comparator): The teeth will undergo a thorough cleaning process using a polishing brush without any paste, and the surfaces will be subsequently air-dried. The application of a single dose of Bifluorid 10 (by VOCO) will be carried out using a micro brush. A thin coat of varnish will be applied to the tooth surface, and it will be left in place for 10-20 seconds before being air-dried. This procedure is designed to facilitate the effective application of the desensitizing agent.
  Interventions: Drug: Fluoride varnish

INTERVENTIONS:
Drug: Gluma Desensitizer — Each sensitive tooth will be cleaned with a polishing paste, rinsed with water and air dried. Two coats of Gluma Desensitizer will be applied using a disposable brush applicator following the manufacturer's instructions and left untouched for 30-60 minutes.
  Arms: Combination of Gluma and Bioactive glass; Gluma Group
Drug: Bioactive glass — The NSK Prophymate Neo will be utilized to dispense Sylc dry powder, which comprises calcium sodium phosphosilicate, onto the sensitive areas. The air stream will be carefully adjusted to 40-46 psi in accordance with the manufacturer's instructions. The handpiece will be maintained at a constant distance of 3-4 mm from the tooth surface, positioned at 60-80 degrees on the buccal surfaces. The powder will be applied for 5-10 seconds per tooth, using a circular motion.
  Other Names: Sylc
  Arms: Bioactive Glass Group; Combination of Gluma and Bioactive glass
Drug: Fluoride varnish — The application of a single dose of Bifluorid 10 (by VOCO) will be carried out using a micro brush. A thin coat of varnish will be applied to the tooth surface, and it will be left in place for 10-20 seconds before being air-dried.
  Other Names: Bifluorid 10
  Arms: Fluoride Varnish

SUMMARY:
Type of study: (A Randomized Controlled Clinical Trial)

Aim :The aim of this randomized controlled clinical trial is to evaluate the effect of Gluma, Bioactive Glass and combination of both, compared to Flouride Varnish on the treatment of dentin hypersensitivity of cervical non-carious lesions in adult Population over six months.

The study will enroll 40 patients meeting the inclusion criteria. Each patient will contribute one tooth with complaints that meet the inclusion criteria, resulting in a total of 40 included teeth. The teeth will be categorized into Four groups based on the type of desensitizer used.

* Group 1 (G1); patients will be randomly assigned to Gluma.
* Group 2 (G2); patients will be randomly assigned to Bioactive Glass Powder.
* Group 3 (G3); patients will be randomly assigned to combination of both materials, Gluma and Bioactive Glass powder
* Group 4 (G4); patients will be randomly assigned to the Fluoride Varnish. For each patient, a sensitivity test will be conducted using a Visual Analog Scale immediately after desensitizer application, as well as at three months and six months post-application.

Clinical procedures:

The study will involve applying a controlled air stimulus (evaporative) to the complaining tooth. This will be done using a dental syringe adjusted to 40-65 psi, directed perpendicular at a distance of 1-3 mm from the exposed dentin. Subsequently, the patient will indicate the level of sensitivity on a Visual Analog Scale (VAS) chart ranging from 0 to 10, with a focus on instances where the VAS score exceeds 4. To facilitate the patient's expression of pain intensity, a plastic card featuring figures with facial expressions, color-coded, and numbered, will be utilized. This visual aid aims to streamline the process of discerning and recording the degree of pain experienced by the patient.

For Gluma group

Each sensitive tooth will be cleaned with a polishing paste, rinsed with water and air dried. Two coats of Gluma Desensitizer will be applied using a disposable brush applicator following the manufacturer's instructions and left untouched for 30-60 minutes.

For Bioactive Glass group :

To maintain a dry and clear field of vision, cheek retractors and high-volume suction will be employed during the procedure. High-volume suction, featuring a 45-degree beveled end, will be strategically positioned at the incisal or occlusal part of the teeth. This placement is designed to efficiently remove any particles, preventing the patient from swallowing them and minimizing the risk of minor injuries resulting from a forceful powder and water stream. The NSK Prophymate Neo will be utilized to dispense Sylc dry powder, which comprises calcium sodium phosphosilicate, onto the sensitive areas. The air stream will be carefully adjusted to 40-46 psi in accordance with the manufacturer's instructions. The handpiece will be maintained at a constant distance of 3-4 mm from the tooth surface, positioned at 60-80 degrees on the buccal surfaces. To prevent gingival injury, the tip of the handpiece will be directed incisally during application. The powder will be applied for 5-10 seconds per tooth, using a circular motion.

For the combined group (Bioactive Glass + Gluma) A combination of both Gluma and bioactive glass powder will be applied to the assigned teeth.

For the comparator group :

The teeth will undergo a thorough cleaning process using a polishing brush without any paste, and the surfaces will be subsequently air-dried. The application of a single dose of Bifluorid 10 (by VOCO) will be carried out using a micro brush. A thin coat of varnish will be applied to the tooth surface, and it will be left in place for 10-20 seconds before being air-dried. This procedure is designed to facilitate the effective application of the desensitizing agent.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age ranges from 21- 40 years old.
2. Males or Females
3. Co-operative Patients approving the trial.
4. Good oral hygiene
5. Not received antibiotic therapy for 1 month before sampling

Exclusion Criteria:

1. Lack of compliance
2. Patients with bad oral hygiene
3. Patients who are allergic to any ingredients used in the study.
4. Medically compromised patients with systemic complications that would alter the treatment.
5. Patients who did any periodontal surgeries within the previous 6 months.
6. Inability to give informed consent.
7. Xerostomia.
8. Pregnancy

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Post-operative hypersensitivity assessment using Visaul | From enrollment to the end of treatment at 6 months .
  Post-operative hypersensitivity assessment will be conducted immediately after application, as well as at three months and six months post-treatment. The evaluation will utilize the Visual Analog Scale (VAS) as described by Van den Breemer et al. (2019) . This scale is represented by a horizontal line graded from 1 to 10, with a descriptor at its far-left end indicating no pain and at its far-right end indicating the worst possible pain. Additionally, facial expressions with color codes will be illustrated below the 10-centimeter line on the Visual Analog Scale, as outlined by Burrow et al. (2009). This approach provides a comprehensive and visual means for patients to express and quantify their post-operative hypersensitivity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Elshorouk City, Egypt